CLINICAL TRIAL: NCT02618850
Title: Study of the Role of Metabolic Response Measured by PET/CT Scan After 1 Cycle of First-line Therapy in Patients With Advanced Colorectal Cancer (CRC)
Brief Title: PET/CT Scan as a Tool to Rationalize the Treatment of Patients With Advanced ColoRectal Cancer Undergoing First-line Medical Treatment
Acronym: PETRA2 - CRC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PETRA2 - CRC
Record Dates: First submitted 2015-04-13; First posted 2015-12-02 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer Stage IV
Keywords: metabolic response; chemotherapy; PET
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Advanced CRC patients undergoing first-line chemotherapy (Other): single cohort
  Interventions: Procedure: PET/CT; Drug: first-line chemotherapy

INTERVENTIONS:
Procedure: PET/CT — PET/CT scan at baseline and 10-14 days after day 1 of first cycle chemotherapy
Drug: first-line chemotherapy — as prescribed by oncologist

SUMMARY:
The purpose of this study is to test whether an early metabolic response, measured by PET/CT scan after the first cycle of chemotherapy, is able to predict which patients with advanced CRC have a better prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis histologically confirmed colorectal carcinoma
* stage IV disease
* patients eligible for standard first-line treatment medical therapy (chemotherapy, and when indicated in association with EGFR inhibitor and/or antiangiogenic) for advanced disease, at diagnosis or after primary surgery.
* At least one target or non-target lesion according to RECIST revised version 1.1.
* Age > or = 18 years .
* ECOG PS 0-2.
* Life expectancy > 3 months.
* Signed informed consent.

Exclusion Criteria:

* Uncontrolled diabetes (glucose > 200 mg/dl
* Any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer or surgically resected prostate cancer with normal PSA).
* Pregnant or lactating females.
* Previous medical therapy for metastatic disease (prior surgery, radiation therapy are permitted, as well as adjuvant medical therapy completed at least 6 months prior to study entry).
* Any poorly controlled illness (including active infections, significant hepatic, renal, metabolic or cardiac disease, myocardial infarction within previous 12 months) that may, according to physician's judgement, interfere with the patient's ability to undergo chemotherapy and/or the examinations within the study protocol
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2014-04; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline in highest value SUVmax (maximum standardized uptake values in PET/CT scan) | 2 weeks
  To validate as prognostic factor, in terms of overall survival,early metabolic response, defined as a reduction of more than 50% of the highest value of SUVmax recorded at PET/CT scan after one cycle of chemotherapy, compared to the highest value of SUVmax recorded baseline examination

SECONDARY OUTCOMES:
Change from baseline in SUVmaxsum, TLGmax and TLGmaxsum | one year
  to describe and validate early metabolic response as a prognostic factor (in terms of progression free survival), using the sum of the SUVmax (SUVmaxsum) , the highest value of TLG (TLGmax), the sum of TLG ( TLGmaxsum).
correlation among SUVmax, SUVmaxsum, TLGmax, TLGsum with progression-free survival after first-line pharmacologic therapy | one year
  prognostic role of early metabolic response (defined according the above reported 4 parameters) in terms of progression free survival after a first line pharmacologic therapy
correlation among SUVmax, SUVmaxsum, TLGmax, TLGsum with objective response | 3 months
  To describe the association between early metabolic response (defined according the above reported 4 parameters) and objective response according RECIST criteria, measured after 3 cycles of chemotherapy
prognostic value of metabolic response (SUVmax, SUVmaxsum, TLGmax, TLGsum) and recist response | one year

OTHER OUTCOMES:
prognostic value of metabolic response (SUVmax, SUVmaxsum, TLGmax, TLGsum) by different cut off values (other than 50% reduction) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Secondo Lastoria, M.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute Naples, Italy; Director Clinical Trials Unit; Ciro Gallo, M.D., Ph.D, Principal Investigator — Second University of Naples, Italy; Chair of Medical Statistics; Luigi Aloj, M.D., Principal Investigator — National Cancer Institute, Naples; Corradina Caracò, M.D., Principal Investigator — National Cancer Institute, Naples; Vincenzo Iaffaioli, M.D., Principal Investigator — National Cancer Institute, Naples; Guglielmo Nasti, M.D., Principal Investigator — National Cancer Institute, Naples; Antonio Avallone, M.D., Principal Investigator — National Cancer Institute, Naples; Giovanni Romano, M.D., Principal Investigator — National Cancer Institute, Naples; Paolo Delrio, M.D., Principal Investigator — National Cancer Institute, Naples; Francesco Izzo, M.D., Principal Investigator — National Cancer Institute, Naples
Locations (1):
- Istituto Nazionale dei Tumori, Napoli, Italy